# **Trial Summary Report**

Date: 05/31/2023

Record Verification Date: 03/17/2023

| Trial Identification | |
|-------------------------------|-------------------|
| Trial Category | Complete |
| Trial Type | Interventional |
| NCI Trial Identifier | NCI-2019-07902 |
| Other Trial Identifiers | |
| Lead Organization Identifier | ADVL18P1 |
| ClinicalTrials.gov Identifier | NCT04203316 |
| DCP Identifier | No Data Available |
| CTEP Identifier | ADVL18P1 |
| CCR Identifier | No Data Available |
| Amendment Number | 4 |
| Amendment Date | 12/15/2022 |

| General Trial Details | 6 |
|---|---|
| Туре | Interventional |
| Official Title | An Open-Label Feasibility Study to Assess the Safety and |
| | Pharmacokinetics of Enasidenib in Pediatric Patients with |
| | Relapsed/Refractory Acute Myeloid Leukemia (R/R-AML) with an |
| | Isocitrate Dehydrogenase-2 (IDH2) Mutation |
| Brief Title | Enasidenib for the Treatment of Relapsed or Refractory Acute |
| | Myeloid Leukemia Patients with an IDH2 Mutation |
| Acronym | No Data Available |
| Brief Summary | |

This trial studies the side effects of enasidenib and to see how well it works in treating patients with acute myeloid leukemia that has come back after treatment (relapsed) or has been difficult to treat with chemotherapy (refractory). Patients must also have a specific genetic change, also called a mutation, in a protein called IDH2. Enasidenib may stop the growth of cancer cells by blocking the mutated IDH2 protein, which is needed for cell growth.

# Detailed Description

# PRIMARY OBJECTIVES:

- I. To determine the safety of treatment with enasidenib mesylate (enasidenib) administered at continuous daily oral dosing for a 28-day cycle up to 12 cycles in pediatric patients with IDH2-mutant relapsed/refractory (R/R)-acute myeloid leukemia (AML).
- II. To characterize the plasma pharmacokinetic (PK) profile of enasidenib in pediatric patients with IDH2-mutant R/R-AML.

# SECONDARY OBJECTIVES:

I. To investigate the pharmacodynamic (PD) relationship of oncogenic metabolite

2-hydroxyglutarate (2-HG) to enasidenib treatment in pediatric patients with IDH2-mutant R/R-AML.

II. To describe the clinical activity of enasidenib in pediatric patients with IDH2-mutant R/R-AML.

# OUTLINE:

Patients receive enasidenib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and/or biopsy and collection of blood on study.

After completion of study treatment, patients are followed up at 30 days, then periodically up to 1 year.

| Sponsor | Children's Oncology Group |
|---|---|
| Lead Organization | Children's Oncology Group |
| Principal Investigator | Zarnegar-Lumley, Sara |
| Responsible Party | Sponsor |
| Overall Official | Zarnegar-Lumley, Sara (Principal Investigator), Children's |
| | Oncology Group |

| Status/Dates | |
|-------------------------|-------------------------|
| Current Trial Status | Active as of 01/30/2023 |
| Trial Start Date | 03/30/2020-Actual |
| Primary Completion Date | 12/31/2030-Anticipated |
| Trial Completion Date | 12/31/2030-Anticipated |

| Regulatory Information | |
|-------------------------------|-------------------|
| Studies a U.S. FDA-regulated | No Data Available |
| Drug Product | |
| Studies a U.S. FDA-regulated | No Data Available |
| Device Product | |
| Product Exported from the U.S | No Data Available |
| FDA Regulated Intervention? | Yes |
| Section 801? | Yes |
| DMC Appointed? | No |
| IND/IDE Study? | Yes |

| Human Subject Safety | |
|-----------------------|---------------------|
| Board Approval Status | Submitted, approved |
| Board Approval Number | 12/15/2022 |

| IND/IDE | | | | | | |
|---|---|---|---|---|---|---|
| Туре | Grantor | Number | Holder Type | Holder | | Expanded<br>Access<br>Record |
| IND | CDER | 146610 | Organization | | Unknown | |

| NIH Grants | | | |
|---|---|---|---|
| Funding Mechanism | NIH Institution Code | | NCI Division/Program<br>Code |
| U10 | CA | 180886 | CTEP |

| Data Table 4 Information | |
|--------------------------------|---------------------------|
| Funding Category | National |
| Funding Sponsor/Source | Children's Oncology Group |
| Anatomic Site Code | |
| Myeloid and Monocytic Leukemia | |

| Collaborators | |
|---------------------------|----------------|
| Name | Role |
| National Cancer Institute | Funding Source |

| Disease/Condition |
|-----------------------------------|
| Name |
| Recurrent Acute Myeloid Leukemia |
| Refractory Acute Myeloid Leukemia |

| Trial Design | |
|----------------------------|-------------------|
| Туре | Interventional |
| Primary Purpose | Treatment |
| Pragmatic Trial | No |
| Phase | II. |
| Pilot Study? | No |
| Interventional Study Model | Single Group |
| Model Description | No Data Available |
| Number of Arms | 1 |
| Masking | No Masking |
| Masking Description | No Data Available |

| Allocation | NA |
|-------------------|----|
| Target Enrollment | 10 |

| Eligibility Criteria | |
|-----------------------------|-----------|
| Accepts Healthy Volunteers? | No |
| Sex | All |
| Minimum Age | 24 Months |
| Maximum Age | 21 Years |

# **Inclusion Criteria**

- Patients must be >= 24 months and < 21 years of age at the time of study enrollment</li>
- Patient must have AML with an IDH2 mutation identified from a peripheral blood or bone marrow sample at the time of diagnosis and/or relapsed/refractory disease
- Patient must have bone marrow assessment (aspiration or biopsy) with > 5% leukemic blasts by morphology and/or flow cytometry in at least one of the following clinical scenarios:
  - \* Second or greater relapse after chemotherapy or hematopoietic stem cell transplant (HSCT)
  - \* Refractory after >= 2 attempts at induction therapy
- Relapsed patients
  - \* Must not have received prior re-induction therapy for this relapse
  - \* Each block of chemotherapy (i.e., cytarabine, daunorubicin and etoposide [ADE], cytarabine and mitoxantrone [MA]) is a separate re-induction attempt
  - \* Donor lymphocyte infusion (DLI) is considered a re-induction attempt
- Refractory patients
  - \* Each attempt at induction therapy may include up to two chemotherapy courses
- Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
- Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
- Evaluation of cerebrospinal fluid (CSF) is only required if there is a clinical suspicion of central
  nervous system (CNS) involvement by leukemia during eligibility screening. Should a patient be
  found to have CNS2 or CNS3 status by CSF prior to eligibility screening, patient may receive
  intrathecal chemotherapy > 72 hours prior to starting study drug. CNS1 status must be
  established before starting study drug
- Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy
  and must meet the following minimum duration from prior anti-cancer directed therapy prior to
  enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g., blood
  count criteria, the patient is considered to have recovered adequately
  - \* Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
  - \*\* >= 14 days must have elapsed after the completion of other cytotoxic therapy with the exception of hydroxyurea. Additionally, patients must have fully recovered from all acute toxic effects of prior therapy. NOTE: Cytoreduction with hydroxyurea must be discontinued >= 24 hours prior to the start of protocol therapy
  - \*\* Intrathecal chemotherapy must be completed >= 72 hours prior to the start of the first cycle of treatment
  - \* Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment

- \* Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
- \* Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
- \* Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study research coordinator
- \* Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
- \* Stem cell Infusions (with or without total body irradiation [TBI]):
- \*\* Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion:
- \*\*\* >= 60 days after infusion for bone marrow or stem cell transplant and
- \*\*\* >= 4 weeks after infusion for any stem cell infusion including DLI or boost infusion
- \*\*\* There must be no evidence of graft versus host disease (GVHD)
- \*\* Autologous stem cell infusion including boost infusion: >= 42 days
- \* Cellular Therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
- \* XRT/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
- \* Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-metaiodobenzylguanidine [MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
- \* Study-specific limitations on prior therapy: small molecule investigational agents: >= 14 days or > 5 half-lives must have elapsed from the last dose of the agent, whichever is greater
- Platelet count >= 20,000/mm<sup>3</sup> (may receive platelet transfusions)
- Hemoglobin >= 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions)
- Creatinine clearance or radioisotope glomerular filtration rate [GFR] >= 70 ml/min/1.73 m<sup>2</sup> or a serum creatinine based on age/gender as follows:
  - \* Age: Maximum serum creatinine (mg/dL)
  - \*\* 2 to < 6 years: 0.8 (male and female)
  - \*\* 6 to < 10 years: 1 (male and female)
  - \*\* 10 to < 13 years: 1.2 (male and female)
  - \*\* 13 to < 16 years: 1.5 (male); 1.4 (female)
  - \*\* >= 16 years: 1.7 (male); 1.4 (female)
- Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age</li>
- Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 225 U/L.</li>
   For the purpose of this study, the ULN for SGPT is 45 U/L
- Serum albumin >= 2 g/dL
- Left ventricular ejection fraction of >= 50% by echocardiogram
- Regulatory Requirements
  - \* All patients and/or their parents or legal authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines
  - \* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

# **Exclusion Criteria**

- AML associated with Down syndrome or t(15;17) is not eligible for study
- Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained

in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy and for 2 months after the last dose of enasidenib. Abstinence is an acceptable method of birth control. It is not known if enasidenib is present in breast milk. Breastfeeding is not recommended during therapy or for at least 30 days after the last dose of enasidenib

- Concomitant Medications:
  - \* Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid. The use of corticosteroids to manage the side effect of IDH inhibitor-associated differentiation syndrome (IDH-DS), is permitted on study
  - \* Investigational drugs: Patients who are currently receiving another investigational drug are not eligible
  - \* Anti-cancer agents: Patients who are currently receiving other anti-cancer agents are not eligible (except leukemia patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy; the use of hydroxyurea to manage the side effect of IDH-DS, is permitted on study)
  - \* Anti-GVHD agents post-transplant: Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
- Patients must be able to swallow intact tablets whole or use the alternate enasidenib formulation.
  - \* Patients with known hypersensitivity to any of the components of enasidenib are not eligible.
  - \* Patients with prior exposure to enasidenib or another IDH2 inhibitor are not eligible.
  - \* Patients taking the following drugs will be excluded from study entry unless these drugs are discontinued or patients are transferred to a medically acceptable alternative > 5 half-lives before the first dose of enasidenib.
  - \*\* Drugs with a narrow therapeutic range that are sensitive substrates of the following cytochrome P450 (CYP) enzymes: CYP2C8 (e.g. paclitaxel), 2C9 (e.g. phenytoin and warfarin), 2C19 (e.g. s-mephenytoin), 2D6 (e.g. thioridazine), and 1A2 (e.g. theophylline and tizanidine).
  - \*\* Breast cancer resistant protein (BCRP) transporter-sensitive substrate rosuvastatin
- Patients with the following leukemia complications are not eligible for this trial:
  - \* No intrathecal chemotherapy is permitted on study. Prior to study enrollment, cerebrospinal fluid (CSF) evaluation is only required if there is a clinical suspicion for CNS leukemia. Clinical signs of CNS leukemia (such as facial nerve palsy, brain/eye involvement or hypothalamic syndrome) are not eligible for this trial
  - \* Immediately life-threatening, severe complications of leukemia including uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
- Patients who have received a prior solid organ transplantation are not eligible
- Infection: Patients who have an uncontrolled infection or patients with known human immunodeficiency virus (HIV) or active hepatitis B or C are not eligible
- Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

| Intervention(s) | | | |
|---|---|---|---|
| Type | Name | Alternate Name | Description |
| Drug | | 1446502-11-9, AG-221,<br>CC-90007 Free Base, | Given PO |
| | | ENASIDENIB | |
| Drug | Enasidenib Mesylate | 1650550-25-6, | Given PO |

| | | 2-Methyl-1-[(4-[6-(trifluo romethyl)pyridin-2-yl]-6-{[2-(trifluoromethyl)pyridin-4-yl]amino}-1,3,5-tria zin-2-yl)amino]propan-2-ol Methanesulfonate, 2-Propanol, 2-Methyl-1-((4-(6-(trifluo romethyl)-2-pyridinyl)-6-((2-(trifluoromethyl)-4-pyridinyl)amino)-1,3,5-triazin-2-yl)amino)-, Methanesulfonate (1:1), AG-221 Mesylate, CC-90007, ENASIDENIB MESYLATE, Enasidenib Methanesulfonate, Idhifa | |
|---|---|---|---|
| Procedure/Surgery | Bone Marrow Aspiration | Bone Marrow<br>Aspiration, bone<br>marrow aspiration | Undergo bone marrow aspiration |
| Procedure/Surgery | Bone Marrow Biopsy | Biopsy of Bone Marrow,<br>Biopsy, Bone Marrow,<br>bone marrow biopsy,<br>Bone Marrow Biopsy | Undergo bone marrow<br>biopsy |
| Procedure/Surgery | Biospecimen Collection | Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection | Undergo collection of<br>blood |

| Arm/Group(s) | |
|---|---|
| Туре | Experimental |
| Label | Treatment (enasidenib) |
| Description | Patients receive enasidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and/or biopsy and collection of blood on study. |
| Intervention(s) | |

| Туре | Name | Alternate Name | Description |
|---|---|---|---|
| Drug | Enasidenib | 1446502-11-9, AG-221,<br>CC-90007 Free Base,<br>ENASIDENIB | Given PO |
| Drug | Enasidenib Mesylate | 2-Methyl-1-[(4-[6-(trifluo romethyl)pyridin-2-yl]-6-{[2-(trifluoromethyl)pyrid in-4-yl]amino}-1,3,5-tria zin-2-yl)amino]propan-2-ol Methanesulfonate, 2-Propanol, 2-Methyl-1-((4-(6-(trifluo romethyl)-2-pyridinyl)-6-((2-(trifluoromethyl)-4-pyridinyl)amino)-1,3,5-triaz in-2-yl)amino)-, Methanesulfonate (1:1), AG-221 Mesylate, CC-90007, ENASIDENIB MESYLATE, Enasidenib Methanesulfonate, Idhifa | |
| Procedure/Surgery | Bone Marrow Aspiration | | Undergo bone marrow aspiration |
| Procedure/Surgery | Bone Marrow Biopsy | Biopsy of Bone Marrow,<br>Biopsy, Bone Marrow,<br>bone marrow biopsy,<br>Bone Marrow Biopsy | Undergo bone marrow<br>biopsy |
| Procedure/Surgery | Biospecimen Collection | • | Undergo collection of blood |

| Primary Outcome Measures | | |
|---|---|---|
| Title | Description | Time Frame |
| toxicities of enasidenib | Frequencies (%) of patients with a dose limiting toxicity stratified by dose level. | • |
| Area under the plasma | A descriptive analysis of the | Up to 120 days |

| concentration versus time curve of enasidenib | area under the plasma concentration versus time curve of enasidenib including median, minimum and maximum by dose level. | |
|---|---|---|
| Total plasma clearance of enasidenib | A descriptive analysis of the total plasma clearance of enasidenib including median, minimum and maximum by dose level. | Up to 120 days |
| Elimination half-life of enasidenib | A descriptive analysis of the elimination half-life of enasidenib including median, minimum and maximum by dose level. | Up to 120 days |
| Maximum concentration of enasidenib | A descriptive analysis of the maximum concentration of enasidenib including median, minimum and maximum by dose level. | Up to 120 days |

| Secondary Outcome Measures | | |
|---|---|---|
| Title | Description | Time Frame |
| Plasma 2-HG levels of enasidenib | A descriptive analysis of the plasma 2-HG levels of enasidenib including median, minimum and maximum by dose level. | Up to 120 days |
| Overall Response Rate of enasidenib | Frequency (%) of patients with at least partial response by dose level. | Up to 2 years |
| · | frequency of response (%) for | Up to 1 year after last dose of study drug |
| Time to response of enasidenib | 95% confidence interval. | From the date of first dose to the date of first documented response, assessed up to 1 year after last dose of study drug |
| Time to complete remission of enasidenib | 95% confidence interval. | From the date of first dose to the date of first documented CR, assessed up to 1 year after last dose of study drug |
| Duration of response of enasidenib | | From the date of first documented response to the |

| | | date of first documented confirmed disease progression/relapse, or death, whichever occurs first, assessed up to 1 year |
|---|---|---|
| Duration of complete response of enasidenib | Median duration of remission with 95% confidence interval. | From the date of first documented CR to the date of first documented confirmed disease progression/relapse, or death, whichever occurs first, assessed up to 1 year after last dose of study drug |
| Event-free survival of enasidenib | Median time to event with 95% confidence interval. | From the date of first dose to the date of documented confirmed disease progression/relapse, or death, whichever occurs first, assessed up to 1 year after last dose of study drug |
| Overall survival of enasidenib | Median time to death with 95% confidence interval. | From the patient's first dose to the date of the death, or the last date the patient was known to be alive, assessed up to 1 year after last dose of study drug |

| Markers | | | | | |
|---|---|---|---|---|---|
| Marker Name | Evaluation Type | Assay Type | Biomarker Use | Biomarker<br>Purpose | Specimen Type |
| 2-HG (2HG; 2-HG; Alpha-Hydroxyg lutarate; 2-Hydroxypenta nedioic Acid; Alpha-Hydroxyg lutaric Acid; Pentanedioic Acid, 2-Hydroxy-; 2-Hydroxyglutar ic Acid; 2-Hydroxyglutar ate; 2-Hydroxy-Pent anedioic Acid) | | Unspecified | Integrated | Response<br>Assessment | Blood |
| Blasts 5-25 | Level/Quantity | Unspecified | Integrated | Response | Bone Marrow |

| _ | | | | | |
|---|---|---|---|---|---|
| Percent of Bone Marrow | | | | Assessment | |
| Nucleated Cells | | | | | |
| Blasts More<br>than 5 Percent<br>of Bone Marrow<br>Nucleated Cells<br>(Blasts Greater<br>than 5 Percent<br>of Bone Marrow<br>Nucleated<br>Cells; Blasts<br>Over 5 Percent<br>of Bone Marrow<br>Nucleated<br>Cells) | | Flow Cytometry | Integral | Eligibility<br>Criterion -<br>Inclusion | Bone Marrow |
| Blasts Under 5 Percent of Bone Marrow Nucleated Cells (Blasts Less than 5 Percent of Bone Marrow Nucleated Cells) | • | Unspecified | Integrated | Response<br>Assessment | Bone Marrow |
| Bone Marrow Blasts Decreased by 50 Percent or More Compared to Pretreatment Level (Decrease of Pretreatment Bone Marrow Blast Percentage by at Least 50 Percent; Decrease of Pretreatment Bone Marrow Blast Percentage by at Least 50 | Level/Quantity | Unspecified | Integrated | Response<br>Assessment | Bone Marrow |
| IDH2 Gene | Genetic | Unspecified | Integral | Eligibility | Blood, Bone |
| <u> </u> | | • | | | |

| Mutation | Analysis | Criterion - | Marrow |
|----------------|----------|-------------|--------|
| (Isocitrate | | Inclusion | |
| Dehydrogenase | | | |
| (NADP(+)) 2, | | | |
| Mitochondrial | | | |
| Gene Mutation; | | | |
| IDH2 Mutation; | | | |
| Isocitrate | | | |
| Dehydrogenase | | | |
| 1 (NADP+), | | | |
| Mitochondrial | | | |
| Gene Mutation) | | | |

| Participating Sites | | | | |
|---|---|---|---|---|
| PO ID | Facility | Contact | Recruitment Status & Date(s) | Investigator(s) |
| 66945 | Alfred I duPont<br>Hospital for<br>Children,<br>Wilmington, DE<br>19803 USA | Site Public<br>Contact, email:<br>Allison.bruce@ne<br>mours.org, phone:<br>302-651-5572 | Active as of<br>02/01/2023 | <ul> <li>Scott Bradfield -<br/>Principal<br/>Investigator</li> </ul> |
| 29135 | Arkansas<br>Children's Hospital,<br>Little Rock, AR<br>72202-3591 USA | Site Public<br>Contact, email: ,<br>phone:<br>501-364-7373 | Active as of 02/01/2023 | <ul> <li>David Becton -<br/>Principal<br/>Investigator</li> </ul> |
| 133247 | C S Mott Children's<br>Hospital, Ann<br>Arbor, MI 48109<br>USA | Site Public<br>Contact, email: ,<br>phone:<br>800-865-1125 | Active as of 02/01/2023 | <ul> <li>Rajen Mody -<br/>Principal<br/>Investigator</li> </ul> |
| 9858 | Universitaire | Site Public<br>Contact, email:<br>yvan.samson@um<br>ontreal.ca, phone:<br>514-345-4931 | Temporarily<br>Closed to Accrual<br>as of 08/31/2022 | <ul> <li>Yvan Samson -<br/>Principal<br/>Investigator</li> </ul> |
| 58509 | Children's Hospital<br>Colorado, Aurora,<br>CO 80045 USA | Site Public<br>Contact, email:<br>josh.b.gordon@ns<br>mtp.kp.org, phone:<br>303-764-5056 | Active as of 02/01/2023 | <ul> <li>Margaret Macy -<br/>Principal<br/>Investigator</li> </ul> |
| 25745 | Children's Hospital<br>of Alabama,<br>Birmingham, AL<br>35233 USA | Site Public<br>Contact, email:<br>oncologyresearch<br>@peds.uab.edu,<br>phone:<br>205-638-9285 | Active as of 02/01/2023 | <ul> <li>Matthew Kutny -<br/>Principal<br/>Investigator</li> </ul> |

| 196933 | UPMC, Pittsburgh, | Site Public<br>Contact, email:<br>jean.tersak@chp.e<br>du, phone:<br>412-692-8570 | Active as of<br>02/01/2023 | <ul> <li>Andrew Bukowinski - Principal Investigator </li> </ul> |
|---|---|---|---|---|
| 230502 | Children's Hospital<br>of San Antonio,<br>San Antonio, TX<br>78207 USA | Site Public<br>Contact, email:<br>bridget.medina@c<br>hristushealth.org,<br>phone:<br>210-704-2894 | Active as of<br>05/16/2023 | Timothy Griffin - Principal Investigator |
| 238382 | Daughters, Norfolk, | Contact, email: | Active as of<br>02/01/2023 | • Eric Lowe -<br>Principal<br>Investigator |
| 141741 | Children's Mercy<br>Hospitals and<br>Clinics, Kansas<br>City, MO 64108<br>USA | Site Public<br>Contact, email:<br>rryan@cmh.edu,<br>phone:<br>816-302-6808 | Active as of<br>02/01/2023 | <ul> <li>Kevin Ginn -<br/>Principal<br/>Investigator</li> </ul> |
| 65938 | Children's National<br>Medical Center,<br>Washington, DC<br>20010 USA | Site Public<br>Contact, email: ,<br>phone:<br>202-884-2549 | Active as of<br>02/01/2023 | <ul> <li>AeRang Kim -<br/>Principal<br/>Investigator</li> </ul> |
| 182911 | Children's Hospital | Site Public<br>Contact, email:<br>cancer@cchmc.org<br>, phone:<br>513-636-2799 | Active as of<br>02/01/2023 | <ul> <li>Joseph Pressey -<br/>Principal<br/>Investigator</li> </ul> |
| 160485 | Hackensack<br>University Medical<br>Center,<br>Hackensack, NJ<br>07601 USA | Site Public<br>Contact, email: ,<br>phone:<br>201-996-2879 | Active as of<br>02/01/2023 | <ul> <li>Jing Chen - Principal Investigator </li> </ul> |
| 125217 | Kimmel Cancer<br>Center, Baltimore, | Site Public<br>Contact, email:<br>jhcccro@jhmi.edu,<br>phone:<br>410-955-8804 | Active as of<br>02/01/2023 | Alan Friedman - Principal Investigator |
| 65850 | MedStar<br>Georgetown<br>University Hospital,<br>Washington, DC<br>20007 USA | Site Public<br>Contact, email: , | Closed to Accrual<br>as of 11/17/2022 | Nina Kadan-Lottick - Principal Investigator |
| 71176 | Nicklaus Children's<br>Hospital, Miami, FL | | Active as of<br>05/30/2023 | • Ziad Khatib -<br>Principal |

| | 33155 USA | phone:<br>888-624-2778 | | Investigator |
|---|---|---|---|---|
| 105447 | Children,<br>Indianapolis, IN | Site Public<br>Contact, email: ,<br>phone:<br>800-248-1199 | Active as of<br>02/01/2023 | Sandeep Batra - Principal Investigator |
| 60830 | Children-Presbyteri | Site Public<br>Contact, email: ,<br>phone:<br>303-839-6000 | Active as of<br>02/01/2023 | Jennifer Clark - Principal Investigator |
| 221716 | Research Hospital,<br>Memphis, TN | Site Public<br>Contact, email:<br>referralinfo@stjude<br>.org, phone:<br>888-226-4343 | Active as of<br>02/01/2023 | <ul> <li>Jeffrey Rubnitz -<br/>Principal<br/>Investigator</li> </ul> |
| 173533 | New York Upstate<br>Medical University, | Site Public<br>Contact, email: ,<br>phone:<br>315-464-5476 | Active as of<br>02/01/2023 | Philip Monteleone - Principal Investigator |
| 70710 | Science Center -<br>Gainesville, | Site Public<br>Contact, email:<br>cancer-center@ufl.<br>edu, phone:<br>352-273-8010 | Closed to Accrual<br>as of 02/01/2023 | William Slayton - Principal Investigator |
| 190601 | Oklahoma Health<br>Sciences Center,<br>Oklahoma City, OK | Site Public<br>Contact, email:<br>ou-clinical-trials@o<br>uhsc.edu, phone:<br>405-271-8777 | Active as of<br>02/21/2023 | Rene McNall-Knapp - Principal Investigator |
| 226789 | UT<br>Southwestern/Sim<br>mons Cancer<br>Center-Dallas,<br>Dallas, TX 75390<br>USA | Site Public<br>Contact, email:<br>canceranswerline<br>@UTSouthwestern<br>.edu, phone:<br>214-648-7097 | Active as of<br>02/01/2023 | <ul> <li>Kathleen (Wiertel) Ludwig - Principal Investigator</li> </ul> |
| 221306 | Cancer Center, | Site Public<br>Contact, email: ,<br>phone:<br>800-811-8480 | Active as of<br>02/01/2023 | <ul><li>Sara Zarnegar-Lumley - Principal Investigator</li></ul> |